CLINICAL TRIAL: NCT02973087
Title: A PROSPECTIVE, PHASE 3, OPEN-LABEL, INTERNATIONAL MULTICENTER STUDY ON EFFICACY AND SAFETY OF PROPHYLAXIS WITH rVWF IN SEVERE VON WILLEBRAND DISEASE
Brief Title: rVWF IN PROPHYLAXIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 071301; 2016-001478-14 (EudraCT Number)
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases | interventions — von Willebrand Factor; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Study Participants (Experimental): Participants will receive prophylaxis with rVWF in two cohorts: on-demand (OD) cohort (previously treated with OD) and pdVWF switch cohort (participants switching from prophylactic treatment with pdVWF).
  Interventions: Biological: von Willebrand factor (Recombinant); Biological: Antihemophilic Factor (Recombinant)

INTERVENTIONS:
Biological: von Willebrand factor (Recombinant) — OD participants will receive intravenous (IV) rVWF:RCo at an initial prophylactic dose of 50 +/- 10 International Unit per Kilogram (IU/kg) twice (two infusions) a week for at least 12 months up to 15 months and may be increased up to 80 IU/kg. pdVWF switch cohort participants will receive rVWF:RCo equivalent (± 10%) to the weekly VWF dose received during prophylactic treatment with pdVWF.
  Other Names: BAX 111; rVWF; VONVENDI; vonicog alfa; BAX111
Biological: Antihemophilic Factor (Recombinant) — During prophylaxis period any bleeding episodes requiring substitution therapy with VWF concentrate to control bleeding will be treated with rVWF with or without ADVATE. Participants will receive rFVIII IV if necessary for OD treatment of breakthrough bleeds or for peri-operative. The dose will be according to the bleeding type and severity and it will be adjusted to the clinical response.
  Other Names: ADVATE; Recombinant Factor VIII; rFVIII

SUMMARY:
The purpose of this phase 3 study is to investigate the efficacy and safety, including immunogenicity, thrombogenicity and hypersensitivity reactions, as well as pharmacokinetics (PK), health related quality of life (HRQoL) and pharmacoeconomics of prophylactic treatment with recombinant von Willebrand factor (rVWF) (vonicog alfa) in adult participants with severe von Willebrand disease (VWD).

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a documented diagnosis of severe von Willebrand disease (VWD) (baseline Von Willebrand factor: Ristocetin cofactor activity (VWF:RCo) less than (<) 20 International Units/Deciliter [IU/dL]) with a history of requiring substitution therapy with von Willebrand factor concentrate to control bleeding

   1. Type 1 (VWF:RCo <20 IU/dL) or,
   2. Type 2A (as verified by multimer pattern), Type 2B (as diagnosed by genotype), Type 2M or,
   3. Type 3 (Von Willebrand factor antigen (VWF:Ag) less than or equal to [< or =] 3 IU/dL).
2. Diagnosis is confirmed by genetic testing and multimer analysis, documented in patient history or at screening.
3. For on-demand patient group, participant currently receiving on-demand treatment for whom prophylactic treatment is recommended by the investigator.
4. For Plasma derived von Willebrand factor (pdVWF) product switch patient group, participant has been receiving prophylactic treatment of pdVWF products for no less than 12 months prior to screening.
5. For on-demand patient group, participant has greater than or equal to (>or=) 3 documented spontaneous bleeds (not including menorrhagia) requiring von Willebrand factor (VWF) treatment during the past 12 months.
6. Availability of records to reliably evaluate type, frequency and treatment of bleeding episodes during at least 12 months preceding enrollment. Up to 24 months retrospective data should be collected if available. Availability of dosing and factor consumption during 12 months (up to 24 months) of treatment prior to enrollment is required for pdVWF switch participants and is desired (but not a requirement) for on-demand participants.
7. Participant is > or = 18 years old at the time of screening and has a body mass index > or = 15 but <40 kilogram per meter square (kg/m^2).
8. If female of childbearing potential, participant presents with a negative blood/urine pregnancy test at screening and agrees to employ adequate birth control measures for the duration of the study.
9. Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. The participant has been diagnosed with Type 2N Von Willebrand disease (VWD), pseudo VWD, or another hereditary or acquired coagulation disorder other than VWD (eg qualitative and quantitative platelet disorders or prothrombin time [PT]/international normalized ratio [INR] greater than [>]1.4).
2. The participant is currently receiving prophylactic treatment with more than 5 infusions per week.
3. The participant is currently receiving prophylactic treatment with a weekly dose exceeding 240 IU/kg.
4. The participant has a history or presence of a VWF inhibitor at screening.
5. The participant has a history or presence of a Factor VIII (FVIII) inhibitor with a titer ≥0.4 Bethesda units (BU) (by Nijmegen modified Bethesda assay) or > or = 0.6 Bethesda Unit (BU) (by Bethesda assay).
6. The participant has a known hypersensitivity to any of the components of the study drugs, such as to mouse or hamster proteins.
7. The participant has a medical history of immunological disorders, excluding seasonal allergic rhinitis/conjunctivitis, mild asthma, food allergies or animal allergies.
8. The participant has a medical history of a thromboembolic event.
9. The participant is human immunodeficiency virus (HIV) positive with an absolute Helper T cell (CD4) count <200/ cubic millimeter (mm^3).
10. The participant has been diagnosed with significant liver disease per investigator's medical assessment of the participant's current condition or medical history or as evidenced by any of the following: serum alanine aminotransferase (ALT) greater than 5 times the upper limit of normal; hypoalbuminemia; portal vein hypertension (e.g., presence of otherwise unexplained splenomegaly, history of esophageal varices).
11. The participant has been diagnosed with renal disease, with a serum creatinine (CR) level > or = 2.5 milligram per deciliter (mg/dL).
12. The participant has a platelet count <100,000/ milliliter (mL) at screening.
13. The participant has been treated with an immunomodulatory drug, excluding topical treatment (e.g., ointments, nasal sprays), within 30 days prior to signing the informed consent.
14. The participant is pregnant or lactating at the time of enrollment.
15. Patient has cervical or uterine conditions causing menorrhagia or metrorrhagia (including infection, dysplasia).
16. The participant has participated in another clinical study involving another Investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
17. The participant has a progressive fatal disease and/or life expectancy of less than 15 months.
18. The participant is scheduled for a surgical intervention.
19. The participant is identified by the investigator as being unable or unwilling to cooperate with study procedures.
20. The participant has a mental condition rendering him/her unable to understand the nature, scope and possible consequences of the study and/or evidence of an uncooperative attitude.
21. The participant is in prison or compulsory detention by regulatory and/or juridical order.
22. The participant is member of the study team or in a dependent relationship with one of the study team members which includes close relatives (i.e., children, partner/spouse, siblings and parents) as well as employees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (33):
- United States (8):
  - University of Colorado Health, Loveland, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Florida College of Medicine, Jacksonville, Florida
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - University of Colorado Health, Aurora, Indiana
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center of Wake Forest Unversity, Winston-Salem, North Carolina
- Hamilton Health Sciences Centre, Hamilton, Canada
- France (5):
  - Hôpital Morvan, Brest, Finistere
  - Groupement Hospitalier Est- Hôpital Louis Pradel, Bron
  - CHU CAEN - Hôpital de la Côte de Nacre, Caen
  - CHU Dijon - Hopital du Bocage, Dijon
  - Hopital Cardiologique - CHU Lille, Lille
- Germany (4):
  - Coagulation Research Centre GmbH, Duisburg
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Werlhof-Institut GmbH, Hanover
  - Medizinische Hochschule Hannover, Hanover
- Italy (5):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Russia (3):
  - SBEI HPE Altai State Medical University of MoH and SD, Barnaul
  - SAIH "Kemerovo Regional Clinical Hospital", Kemerovo
  - FSBI of Science "Kirov Scientific and Research Institute of Hematology and Blood Transfusion of FMBA, Kirov
- Spain (3):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Turkey (Türkiye) (3):
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Ondokuz Mayis Univ. Med. Fac., Samsun

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Hancock JM, Escobar MA. An evaluation of von Willebrand factor (recombinant) therapy for adult patients living with severe type 3 von Willebrand disease. Expert Rev Hematol. 2023 Mar;16(3):157-161. doi: 10.1080/17474086.2023.2184339. Epub 2023 Mar 2. PMID 36861346
- [Derived] Leebeek FWG, Peyvandi F, Escobar M, Tiede A, Castaman G, Wang M, Wynn T, Baptista J, Wang Y, Zhang J, Mellgard B, Ozen G. Recombinant von Willebrand factor prophylaxis in patients with severe von Willebrand disease: phase 3 study results. Blood. 2022 Jul 14;140(2):89-98. doi: 10.1182/blood.2021014810. PMID 35439298
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc34db2bf003ab45955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 32 sites in the United States, Canada, France, Germany, Italy, Netherlands, Russia, Spain, and Turkey between 16 November 2017 (first participant first visit) and 06 July 2020 (last participant last visit).
Pre-assignment Details: A total of 29 participants were screened, out of which 6 participants were screen failures and 23 participants were grouped into 2 cohorts: Prior On-demand and Switch (based on the previous von Willebrand disease [VWD] treatment they received prior to the study) and received prophylactic treatment with recombinant von Willebrand factor (rVWF).
Groups:
- Prior On-demand Participants: Participants who had taken only on-demand von Willebrand factor (VWF) prior to the current study received rVWF (vonicog alpha) initial prophylactic treatment at a dose range of 50 plus minus (+/- ) 10 international unit per kilogram (IU/kg), intravenous infusion, twice per week for a planned period of 12 months. Dose escalation to higher dose (up to 80 IU/kg per infusion) or frequency (up to 3 times a week) was based on medical indication and investigator judgment. During this prophylactic treatment period, any breakthrough bleeding episodes requiring replacement therapy with VWF concentrate was treated with rVWF with or without ADVATE (recombinant Factor VIII [rFVIII]); the dose was determined according to the bleeding type and severity, and was adjusted based on the participant's clinical response.
- Switch Participants: Participants who had taken prophylactic treatment with plasma derived VWF product (pdVWF) prior to current study and switched to prophylaxis with rVWF (vonicog alpha) during the study for a planned period of 12 months; received rVWF twice weekly at an initial prophylactic dose of +/- 10 percent (%) of VWF in the pdVWF weekly dose received prior to this study. Dosing with rVWF up to 80 IU/kg per infusion or at a frequency up to 3 times a week or once a week were allowed depending on the total weekly dose and the dosing regimen used in their previous pdVWF prophylaxis regimen and based on medical indication and investigator judgment. During this prophylactic treatment period, any breakthrough bleeding episodes requiring replacement therapy with VWF concentrate was treated with rVWF with or without ADVATE (rFVIII); the dose was determined according to the bleeding type and severity, and was adjusted based on the participant's clinical response.
Period: Overall Study
Arm/Group | Prior On-demand Participants | Switch Participants
Started | 13 | 10
Completed | 9 | 8
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) composed of all participants who received any amount of investigational product (IP) (rVWF, vonicog alpha).
Groups:
- Prior On-demand Participants: Participants who had taken only on-demand VWF prior to the current study received rVWF (vonicog alpha) initial prophylactic treatment at a dose range of 50 +/- 10 IU/kg, intravenous infusion, twice per week for a planned period of 12 months. Dose escalation to higher dose (up to 80 IU/kg per infusion) or frequency (up to 3 times a week) was based on medical indication and investigator judgment. During this prophylactic treatment period, any breakthrough bleeding episodes requiring replacement therapy with VWF concentrate was treated with rVWF with or without ADVATE (rFVIII); the dose was determined according to the bleeding type and severity, and was adjusted based on the participant's clinical response.
- Switch Participants: Participants who had taken prophylactic treatment with pdVWF prior to current study and switched to prophylaxis with rVWF (vonicog alpha) during the study for a planned period of 12 months; received rVWF twice weekly at an initial prophylactic dose of +/- 10 percent (%) of VWF in the pdVWF weekly dose received prior to this study. Dosing with rVWF up to 80 IU/kg per infusion or at a frequency up to 3 times a week or once a week were allowed depending on the total weekly dose and the dosing regimen used in their previous pdVWF prophylaxis regimen and based on medical indication and investigator judgment. During this prophylactic treatment period, any breakthrough bleeding episodes requiring replacement therapy with VWF concentrate was treated with rVWF with or without ADVATE (rFVIII); the dose was determined according to the bleeding type and severity, and was adjusted based on the participant's clinical response.
- Total: Total of all reporting groups
Arm/Group | Prior On-demand Participants | Switch Participants | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (17.6) | 43.9 (21.8) | 40.6 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 13 | 7 | 20
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 9 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Annualized Bleeding Rate (ABR) for Spontaneous Bleeding Episodes (BEs) (On-study ABR / Historical ABR) Assessed by Investigator During Prophylactic Treatment With rVWF Through Month 12
Description: ABR for treated spontaneous BEs while on prophylactic treatment with rVWF through month 12 of treatment period/observation period (in years), where an observation period = (date of completion/termination - date of first dose + 1)/365.2425. Bleeds occurred at the same anatomical location with the same etiology within 24 hours after onset of the first bleed were considered a single bleed. Bleeding occurred at multiple locations related to the same injury were considered as a single bleeding episode. Historical observation period for historical BEs was 365 days prior to first dose of study drug. On-study observation period started on the day of first administration of study drug and continuing through the date of completion/discontinuation from study. The comparison of the two ABRs (on-study and historical) for spontaneous bleeding episodes (not related to trauma) during prophylactic treatment with rVWF was reported as a ratio of mean ABRs (on-study ABR:historical ABR).
Time Frame: Up to 12 months
Population: Full analysis set (FAS) composed of all participants who received prophylactic IP treatment.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
ratio | 0.085 [0.021 to 0.346] | 0.550 [0.086 to 3.523]

2. Secondary Outcome: Percentage of Prior On-demand Participants Achieved Spontaneous ABR Percent Reduction Success Through Month 12
Description: For prior on-demand participants, spontaneous ABR percent reduction success was defined as at least 25% reduction of the ABR for treated spontaneous (not related to trauma) BEs during the first 12 months of rVWF (vonicog alfa) prophylaxis relative to the participant's own historical treated spontaneous ABR. Percentage of participants with ABR percent reduction success for on-demand cohort was reported.
Time Frame: Up to 12 months
Population: FAS composed of all participants who received prophylactic IP treatment. This outcome measure was analyzed only for prior on-demand participants treated for spontaneous BEs.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 13
percentage of participants | 92.3 [64.0 to 99.8]

3. Secondary Outcome: Percentage of Switch Participants With Spontaneous ABR Preservation Success Through Month 12
Description: For switch participants, spontaneous ABR preservation success was defined as achieving an ABR for treated spontaneous BEs during first 12 months of rVWF (vonicog alfa) prophylaxis that was no greater than the participant's own historical ABR for treated spontaneous BEs during prophylactic treatment with pdVWF. Percentage of participants with ABR preservation success in switch cohort was reported.
Time Frame: Up to 12 months
Population: FAS composed of all participants who received prophylactic IP treatment. This outcome measure was analyzed only for switch participants treated for spontaneous BEs.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Switch Participants
Number analyzed (Participants) | 10
percentage of participants | 90.0 [55.5 to 99.7]

4. Secondary Outcome: Number of Participants Based on Categorized Spontaneous ABR (sABR) Through Month 12
Description: The sABR was the number of spontaneous bleeds divided by the observation period in years, where an observation period = (date of completion/termination-date of first dose+1)/365.2425.sABR was categorized based on number of BEs as 0, greater than (>) 0 through 2,>2 through 5,>5 during the prophylactic treatment with rVWF (vonicog alfa) through 12 months. Bleeding at multiple locations related to the same injury was counted as single bleeding episode. BEs of unknown cause were counted as spontaneous bleeds. Observation period for historical BEs was 365 days prior to first dose of study drug. The baseline sABR for treated BEs was based on historical BE data and on-study sABR was based on treated spontaneous BEs during prophylaxis with rVWF through Month 12. On-study observation period started on the day of first administration of study drug continuing through the date of completion/discontinuation from study. Number of participants based on categorized sABR was calculated and reported.
Time Frame: Baseline through Month 12
Population: FAS composed of all participants who received prophylactic IP treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
Participants
  Historical: 0 BEs | 0 | 6
  Historical: >0 through 2 BEs | 0 | 3
  Historical: >2 through 5 BEs | 10 | 0
  Historical: >5 BEs | 3 | 1
  On-Study Through Month 12: 0 BEs | 11 | 7
  On-Study Through Month 12: >0 through 2 BEs | 0 | 1
  On-Study Through Month 12: >2 through 5 BEs | 1 | 1
  On-Study Through Month 12: >5 BEs | 1 | 1

5. Secondary Outcome: Total Number of Infusions Administered Per Participant During Prophylactic Treatment With rVWF Through Month 12
Description: For each participant, the total number of infusions was counted as the total number of unique infusions of rVWF which were administered between the dates of informed consent and termination from the study, inclusive, regardless of the date and time of administration. The total number of infusions administered during the study was entered in electronic case record form (eCRF), and recorded in ERT system. Total number of infusions administered per participant during prophylactic treatment With rVWF through 12 months was calculated.
Time Frame: Up to 12 months
Population: FAS composed of all participants who received prophylactic IP treatment.
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
infusions | 65.1 (38.4) | 87.8 (30.2)

6. Secondary Outcome: Average Number of Infusions Per Week Per Participant During Prophylactic Treatment With rVWF Through Month 12
Description: Average number of infusions per week per participant during prophylactic treatment With rVWF through 12 months was calculated.
Time Frame: Up to 12 months
Population: FAS composed of all participants who received prophylactic IP treatment.
Measure: Mean (Standard Deviation); unit: infusions per week
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
infusions per week | 1.88 (0.7) | 1.85 (0.4)

7. Secondary Outcome: Total Weight Adjusted Consumption of rVWF Per Participant During Prophylactic Treatment Through Month 12
Description: For each participant, the body weight-adjusted dose (IU/kg) was derived as the number of units of rVWF infused (IU) divided by the last available body weight (kilogram [kg]) prior to the infusion. Total weight adjusted consumption of rVWF (vonicog alfa) per participant during prophylactic treatment was reported.
Time Frame: Up to 12 months
Population: FAS composed of all participants who received prophylactic IP treatment.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
IU/kg | 3431.584 (2117.6562) | 4433.752 (1844.8761)

8. Secondary Outcome: Number of Treated Spontaneous BEs by Location of Bleeding While on Prophylactic Treatment With rVWF Through Month 12
Description: Number of treated spontaneous BEs by location of bleeding (for example: oral and other mucosa, menorrhagia, hemarthrosis, etc.) while on prophylactic treatment with rVWF was reported.
Time Frame: Up to 12 months
Population: FAS composed of all participants who received prophylactic IP treatment.
Measure: Number; unit: number of BEs
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
number of BEs
  Oral and other mucosa | 5 | 14
  Menorrhagia | 3 | 0
  Hemarthrosis | 0 | 1
  Other | 1 | 0
  Unknown | 0 | 3

9. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered IP that does not necessarily have a causal relationship with the treatment. TEAEs were events which occurred on or after the date and time of administration of the first dose of study medication. TEAEs included both serious AEs and non-serious AEs. Number of participants with TEAEs and serious TEAEs were reported.
Time Frame: From first dose of study drug up to end of study (approximately 32 months)
Population: SAS composed of all participants who received any amount of IP (rVWF, vonicog alpha).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
Participants
  Participants With TEAEs | 10 | 7
  Participants with serious TEAEs | 1 | 2

10. Secondary Outcome: Number of Participants Based on Severity of TEAEs
Description: An AE is defined as any untoward medical occurrence in a participant administered IP that does not necessarily have a causal relationship with the treatment. TEAEs were events which occurred on or after the date and time of administration of the first dose of study medication. TEAEs included both serious AEs and non-serious AEs. Severity of TEAEs was determined by following definitions: Mild: No limitation of usual activities; Moderate: Some limitation of usual activities and may required therapeutic intervention; Severe: Inability to carry out usual activities with sequelae, which required therapeutic intervention. Participants were counted by considering the maximum severity of TEAEs.
Time Frame: From first dose of study drug up to end of study (approximately 32 months)
Population: SAS composed of all participants who received any amount of IP (rVWF, vonicog alpha).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
Participants
  Mild | 7 | 4
  Moderate | 1 | 2
  Severe | 2 | 1

11. Secondary Outcome: Number of Participants With TEAEs Based Causality
Description: An AE was defined as any untoward medical occurrence in a participant administered IP that does not necessarily have a causal relationship with the treatment. TEAEs were events which occurred on or after the date and time of administration of the first dose of study medication. TEAEs included both serious AEs and non-serious AEs. For each AE, the investigator assessed the causal relationship between the IP and the AE based on clinical expertise and judgment according to the following circumstances of the AE: Not related, Unlikely related, Possibly related, or Probably related. A related TEAE was defined as any TEAE indicated as 'possibly related' or 'probably related'. Number of participants with TEAEs based causality was reported.
Time Frame: From first dose of study drug up to end of study (approximately 32 months)
Population: SAS composed of all participants who received any amount of IP (rVWF, vonicog alpha).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
Participants | 1 | 0

12. Secondary Outcome: Number of Participants With Thromboembolic Events
Description: Thromboembolism defined as formation in a blood vessel of a clot (thrombus) that breaks loose and carried by the blood stream and could plug another vessel. Number of participants with thromboembolic events as TEAEs of special interest was reported. A broad standard search query approach was used (broad SMQ) to identify all potential thromboembolic events of interest which were then medically assessed. Number of participants with thromboembolic events as TEAEs of special interest was reported.
Time Frame: From first dose of study drug up to end of study (approximately 32 months)
Population: SAS composed of all participants who received any amount of IP (rVWF, vonicog alpha).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
Participants | 1 | 0

13. Secondary Outcome: Number of Participants With Hypersensitivity Reactions
Description: Hypersensitivity (also called hypersensitivity reaction or intolerance) defined as undesirable reactions produced by the normal immune system, including allergies and autoimmunity. Potential hypersensitivity events were identified by broad search criteria and then medically assessed. Number of participants with hypersensitivity reactions as TEAEs of special interest was calculated.
Time Frame: From first dose of study drug up to end of study (approximately 32 months)
Population: SAS composed of all participants who received any amount of IP (rVWF, vonicog alpha).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
Participants | 0 | 1

14. Secondary Outcome: Number of Participants Who Developed Neutralizing Antibodies to Von Willebrand Factor (rVWF) and Factor VIII (FVIII)
Description: Three functional VWF assays for von Willebrand factor collagen binding (VWF:CB), von Willebrand factor: Ristocetin Cofactor (VWF:RCo) and von Willebrand factor VIII B (VWF:FVIIIB) were used to test the presence of neutralizing anti-VWF antibodies. Neutralizing antibodies to VWF:RCo, VWF:CB and VWF:FVIIIB activities was measured by assays based on the Bethesda assay established for quantitative analysis of FVIII inhibitors (Nijmegen modification of the Bethesda assay). Only confirmed neutralizing anti -VWF antibodies were considered inhibitors. Number of participants who developed neutralizing antibodies to rVWF and FVIII were assessed.
Time Frame: Baseline through Month 12
Population: SAS composed of all participants who received any amount of IP (rVWF, vonicog alpha).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
Participants | 0 | 0

15. Secondary Outcome: Number of Participants Who Developed of Total Binding Antibodies to Von Willebrand Factor (rVWF) and Factor VIII (FVIII)
Description: The presence of total binding anti-VWF antibodies was determined by an enzyme-linked immunosorbent assay (ELISA) employing polyclonal anti-human Immunoglobulin (Ig) antibodies (IgG, IgM and IgA). Binding antibodies against FVIII was analyzed using a proprietary enzyme immunoassay. Number of participants who developed of total binding antibodies to rVWF and FVIII was assessed.
Time Frame: Baseline through Month 12
Population: SAS composed of all participants who received any amount of IP (rVWF, vonicog alpha).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
Participants | 0 | 0

16. Secondary Outcome: Number of Participants Who Developed Binding Antibodies to Chinese Hamster Ovary (CHO) Proteins, Mouse Immunoglobulin G (IgG) and/or rFurin
Description: Total Ig antibodies (IgG, IgA, IgM) against CHO protein and human furin was analyzed using ELISA. For detection and quantification of IgG antibodies originating from human plasma that were directed against mouse-IgG (HAMA: human anti- mouse antibodies) was assessed using ELISA (Medac, Hamburg, Germany). Number of participants who developed binding antibodies to CHO proteins, Mouse IgG and/or rFurin was assessed.
Time Frame: Baseline through Month 12
Population: SAS composed of all participants who received any amount of IP (rVWF, vonicog alpha).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
Participants | 0 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included blood pressure (systolic and diastolic), pulse rate, respiratory rate and body temperature. Number of participants with clinically significant change from baseline in vital signs was assessed.
Time Frame: Baseline up to end of study (approximately 32 months)
Population: SAS composed of all participants who received any amount of IP (rVWF, vonicog alpha).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
Participants | 0 | 0

18. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included hematology and clinical chemistry assessments. Number of participants with clinically significant change from baseline in clinical laboratory parameters was assessed.
Time Frame: Baseline up to end of study (approximately 32 months)
Population: SAS composed of all participants who received any amount of IP (rVWF, vonicog alpha).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 13 | 10
Participants | 0 | 0

19. Secondary Outcome: Pharmacokinetic (PK) Assessment: Incremental Recovery (IR) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: IR at the maximum plasma concentration of VWF:RCo activity at initial PK assessment was reported. Unit of measure: International Units per deciliter/International Units per kilogram ([IU/dL]/[IU/kg]).
Time Frame: At baseline: Within 30 minutes pre-infusion; and post-infusion at 15, 30 minutes and 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours
Population: PK full analysis set (PKFAS) composed of all participants who received at least one IP infusion and who provided at least one quantifiable pharmacokinetic or pharmacodynamic post dose measurement for pharmacokinetic and/or pharmacodynamics analysis. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure. As planned, this outcome measure was assessed only for prior on-demand participants.
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 11
(IU/dL)/(IU/kg) | 1.463 (0.3205)

20. Secondary Outcome: Pharmacokinetic Assessment: Incremental Recovery (IR) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: IR based on VWF:Ag activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: PKFAS composed of all participants who received at least one IP infusion and who provided at least one quantifiable pharmacokinetic or pharmacodynamic post dose measurement for pharmacokinetic and/or pharmacodynamics analysis. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure. As planned, this outcome measure was assessed only for prior on-demand participants.
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
(IU/dL)/(IU/kg) | 1.699 (0.3488)

21. Secondary Outcome: Pharmacokinetic Assessment: Incremental Recovery (IR) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: IR at the maximum plasma concentration of VWF:CB activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
(IU/dL)/(IU/kg) | 2.405 (0.5737)

22. Secondary Outcome: Pharmacokinetic Assessment: Terminal Half-life (T1/2) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: T1/2 defined as the time in hours required for the concentration of the drug to reach half of its original value. T1/2 based on VWF:Rco activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 11
hours | 15.98 [9.01 to 45.8]

23. Secondary Outcome: Pharmacokinetic Assessment: Terminal Half-life (T1/2) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: T1/2 defined as the time in hours required for the concentration of the drug to reach half of its original value. T1/2 based on VWF:Ag activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
hours | 21.81 [12.6 to 39.3]

24. Secondary Outcome: Pharmacokinetic Assessment: Terminal Half-life (T1/2) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: T1/2 defined as the time in hours required for the concentration of the drug to reach half of its original value. T1/2 based on VWF:CB activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
hours | 18.64 [12.8 to 29.4]

25. Secondary Outcome: Pharmacokinetic Assessment: Mean Residence Time (MRT) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: MRT was calculated as (AUMC0-∞/AUC0-∞) - T1/2 where T1 represented the time duration of infusion, where AUMC represented the area under the first moment curve. MRT based on VWF:Rco activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 11
hours | 23.27 (11.00)

26. Secondary Outcome: Pharmacokinetic Assessment: Mean Residence Time (MRT) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: MRT was calculated as (AUMC0-∞/AUC0-∞) - T1/2 where T1 represented the time duration of infusion, where AUMC represented the area under the first moment curve. MRT based on VWF:Ag activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
hours | 33.55 (9.777)

27. Secondary Outcome: Pharmacokinetic Assessment: Mean Residence Time (MRT) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: MRT was calculated as (AUMC0-∞/AUC0-∞) - T1/2 where T1 represented the time duration of infusion, where AUMC represented the area under the first moment curve. MRT based on VWF:CB activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
hours | 27.39 (6.860)

28. Secondary Outcome: Pharmacokinetic Assessment: Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: AUC0-∞ based on VWF:Rco activity at initial PK assessment was reported. Unit of measure: International Units*hour per deciliter (IU*h/dL).
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 11
IU*h/dL | 1199 (467.8)

29. Secondary Outcome: Pharmacokinetic Assessment: Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: AUC0-∞ based on VWF:Ag activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
IU*h/dL | 2578 (1067)

30. Secondary Outcome: Pharmacokinetic Assessment: Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: AUC0-∞ based on VWF:CB activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
IU*h/dL | 3010 (1221)

31. Secondary Outcome: Pharmacokinetic Assessment: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Last Measurable Concentration (AUC0-tlast) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: AUC0-tlast based on VWF:Rco activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
IU*h/dL | 919.8 (378.4)

32. Secondary Outcome: Pharmacokinetic Assessment: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Last Measurable Concentration (AUC0-tlast) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: AUC0-tlast based on VWF:Ag activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
IU*h/dL | 2357 (848.6)

33. Secondary Outcome: Pharmacokinetic Assessment: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Last Measurable Concentration (AUC0-tlast) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: AUC0-tlast based on VWF:CB activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
IU*h/dL | 2824 (1112)

34. Secondary Outcome: Pharmacokinetic Assessment: Maximum Plasma Concentration (Cmax) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: Cmax based on VWF:Rco at initial PK assessment was reported. Unit of measure: International Units per deciliter (IU/dL).
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
IU/dL | 74.62 (16.09)

35. Secondary Outcome: Pharmacokinetic Assessment: Maximum Plasma Concentration (Cmax) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: Cmax based on VWF:Ag activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
IU/dL | 85.1 (19.2)

36. Secondary Outcome: Pharmacokinetic Assessment: Maximum Plasma Concentration (Cmax) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: Cmax based on VWF:CB activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
IU/dL | 120.74 (29.83)

37. Secondary Outcome: Pharmacokinetic Assessment: Minimum Time to Reach the Maximum Plasma Concentration (Tmax) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: Tmax based on VWF:Rco activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
hours | 0.540 [0.27 to 1.02]

38. Secondary Outcome: Pharmacokinetic Assessment: Minimum Time to Reach the Maximum Plasma Concentration (Tmax) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: Tmax based on VWF:Ag activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
hours | 1 [0.27 to 3.25]

39. Secondary Outcome: Pharmacokinetic Assessment: Minimum Time to Reach the Maximum Plasma Concentration (Tmax) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: Tmax based on VWF:CB activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
hours | 0.500 [0.27 to 1.02]

40. Secondary Outcome: Pharmacokinetic Assessment: Volume of Distribution at Steady State (Vss) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss based on VWF:Rco activity at initial assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: deciliter per kilogram (dL/kg)
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 11
deciliter per kilogram (dL/kg) | 1.052 (0.4981)

41. Secondary Outcome: Pharmacokinetic Assessment: Volume of Distribution at Steady State (Vss) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss based on VWF:Ag activity at initial assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
dL/kg | 0.6860 (0.1556)

42. Secondary Outcome: Pharmacokinetic Assessment: Volume of Distribution at Steady State (Vss) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss based on VWF:CB activity at initial assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
dL/kg | 0.4889 (0.1371)

43. Secondary Outcome: Pharmacokinetic Assessment: Clearance (CL) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body. CL based on VWF:Rco activity at initial PK assessment was reported. Unit of measure: deciliter per kilogram per hour (dL/kg/h).
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: dL/kg/h
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 11
dL/kg/h | 0.04765 (0.01620)

44. Secondary Outcome: Pharmacokinetic Assessment: Clearance (CL) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body. CL based on VWF:Ag activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: dL/kg/h
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
dL/kg/h | 0.02185 (0.006821)

45. Secondary Outcome: Pharmacokinetic Assessment: Clearance (CL) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body. CL based on VWF:CB activity at initial PK assessment was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: dL/kg/h
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
dL/kg/h | 0.01872 (0.005946)

46. Secondary Outcome: Pharmacodynamic (PD) Assessment: Maximum Plasma Concentration (Cmax) Based on Factor VIII Clotting (FVIII:C) Activity
Description: Cmax based on FVIII:C activity at initial PD assessment by the 1-stage clotting assay was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
IU/dL | 90.8 (32.1)

47. Secondary Outcome: Pharmacodynamic Assessment: Minimum Time to Reach the Maximum Plasma Concentration (Tmax) Based on Factor VIII Clotting (FVIII:C) Activity
Description: Tmax based on FVIII:C activity at initial PD assessment by the 1-stage clotting assay was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
hours | 24.055 [11.98 to 46.30]

48. Secondary Outcome: Pharmacodynamic Assessment: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Last Measurable Concentration (AUC0-tlast) Based on Factor VIII Clotting (FVIII:C) Activity
Description: AUC0-tlast based on FVIII:C activity at initial PD assessment by the 1-stage clotting assay was reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Prior On-demand Participants
Number analyzed (Participants) | 12
IU*h/dL | 4949 (2436)

49. Secondary Outcome: Pharmacokinetic Assessment at Steady State: Area Under the Plasma Concentration Versus Time Curve From Time 0 to End of the Partial Dosing Interval (AUC0- Tau;ss) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: AUC0-tau;ss based on VWF:Rco activity at steady state during end of study (Month 12) was reported.
Time Frame: At Month 12: Within 30 minutes pre-infusion; and post-infusion at 15, 30 minutes and 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours
Population: PKFAS composed of all participants who received at least one IP infusion and who provided at least one quantifiable pharmacokinetic or pharmacodynamic post dose measurement for pharmacokinetic and/or pharmacodynamics analysis. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 3
IU*h/dL | 1561 (1298) | 1662 (675.0)

50. Secondary Outcome: Pharmacokinetic Assessment at Steady State: Area Under the Plasma Concentration Versus Time Curve From Time 0 to End of the Partial Dosing Interval (AUC0- Tau;ss) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: AUC0-tau;ss based on VWF:Ag activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 3
IU*h/dL | 2908 (1372) | 3196 (838.0)

51. Secondary Outcome: Pharmacokinetic Assessment at Steady State: Area Under the Plasma Concentration Versus Time Curve From Time 0 to End of the Partial Dosing Interval (AUC0- Tau;ss) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: AUC0-tau;ss based on VWF:CB activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 3
IU*h/dL | 3445 (1914) | 4276 (1471)

52. Secondary Outcome: Pharmacokinetics Assessment at Steady State: Maximum Plasma Concentration During the Partial Dosing Interval at Steady State (Cmax;ss) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: Cmax;ss based on VWF:Rco activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
IU/dL | 92.63 (37.05) | 102.89 (44.74)

53. Secondary Outcome: Pharmacokinetics Assessment at Steady State: Maximum Plasma Concentration During the Partial Dosing Interval at Steady State (Cmax;ss) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: Cmax;ss based on VWF:Ag activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
IU/dL | 108.1 (39.6) | 107.1 (37.4)

54. Secondary Outcome: Pharmacokinetics Assessment at Steady State: Maximum Plasma Concentration During the Partial Dosing Interval at Steady State (Cmax;ss) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: Cmax;ss based on VWF:CB activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
IU/dL | 137.48 (44.97) | 162.19 (60.04)

55. Secondary Outcome: Pharmacokinetics Assessment at Steady State: Minimum Time to Reach the Maximum Plasma Concentration at Steady State (Tmax;ss) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: Tmax;ss based on VWF:Rco activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Median (Full Range); unit: hours
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
hours | 0.330 [0.25 to 1.25] | 0.400 [0.33 to 0.52]

56. Secondary Outcome: Pharmacokinetics Assessment at Steady State: Minimum Time to Reach the Maximum Plasma Concentration at Steady State (Tmax;ss) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: Tmax;ss based on VWF:Ag activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Median (Full Range); unit: hours
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
hours | 0.580 [0.28 to 1.17] | 0.330 [0.23 to 1.17]

57. Secondary Outcome: Pharmacokinetics Assessment at Steady State: Minimum Time to Reach the Maximum Plasma Concentration at Steady State (Tmax;ss) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: Tmax;ss based on VWF:CB activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Median (Full Range); unit: hours
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
hours | 0.420 [0.28 to 3.00] | 0.670 [0.33 to 3.02]

58. Secondary Outcome: Pharmacokinetics Assessment at Steady State: Minimum Plasma Concentration During the Partial Dosing Interval at Steady State (Cmin;ss) Based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) Activity
Description: Cmin;ss based on VWF:Rco activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
IU/dL | NA (NA) — Data not reported as value was below the limit of quantification. | NA (NA) — Data not reported as value was below the limit of quantification.

59. Secondary Outcome: Pharmacokinetics Assessment at Steady State: Minimum Plasma Concentration During the Partial Dosing Interval at Steady State (Cmin;ss) Based on Von Willebrand Factor Antigen (VWF:Ag) Activity
Description: Cmin;ss based on VWF:Rco activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
IU/dL | 6.3 (4.8) | 11.7 (8.9)

60. Secondary Outcome: Pharmacokinetics Assessment at Steady State: Minimum Plasma Concentration During the Partial Dosing Interval at Steady State (Cmin;ss) Based on Von Willebrand Factor Collagen Binding (VWF:CB) Activity
Description: Cmin;ss based on VWF:CB activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
IU/dL | 3.82 (6.86) | 9.94 (8.46)

61. Secondary Outcome: Pharmacodynamic Assessment at Steady State: Area Under the Plasma Concentration Versus Time Curve From Time 0 to End of the Partial Dosing Interval (AUC0- Tau;ss) Based on Factor VIII Clotting (FVIII:C) Activity
Description: AUC0-tau;ss based on FVIII:C activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 3
IU*h/dL | 5984 (2490) | 5836 (1735)

62. Secondary Outcome: Pharmacodynamic Assessment at Steady State: Maximum Plasma Concentration During the Partial Dosing Interval at Steady State (Cmax;ss) Based on Factor VIII Clotting (FVIII:C) Activity
Description: Cmax;ss based on FVIII:C activity was assessed at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
IU/dL | 104.1 (35.1) | 75.7 (37.3)

63. Secondary Outcome: Pharmacodynamic Assessment at Steady State: Minimum Time to Reach the Maximum Plasma Concentration at Steady State (Tmax;ss) Based on Factor VIII Clotting (FVIII:C) Activity
Description: Tmax;ss based on FVIII:C activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Median (Full Range); unit: hours
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
hours | 24.500 [6.17 to 29.27] | 24.070 [1.08 to 30.03]

64. Secondary Outcome: Pharmacodynamic Assessment at Steady State: Minimum Plasma Concentration During the Partial Dosing Interval at Steady State (Cmin;ss) Based on Factor VIII Clotting (FVIII:C) Activity
Description: Cmin;ss based on FVIII:C activity at steady state during end of study (Month 12) was reported.
Time Frame: as for outcome 49
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
IU/dL | 15.8 (8.6) | 22.9 (11.3)

65. Secondary Outcome: Factor VIII (FVIII) Clotting Activity
Description: FVIII clotting activity (FVIII:C) levels was assessed and reported as per pre-specified PK time points at Month 12.
Time Frame: as for outcome 49
Population: FAS will be composed of all participants who receive prophylactic IP treatment. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure and "number analyzed" were participants who were evaluable for the outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Prior On-demand Participants | Switch Participants
Number analyzed (Participants) | 9 | 7
IU/dL
  At pre-dose | 22.1 (23.5) | 28.0 (21.2)
  15 minutes post-dose | 28.7 (22.5) | 30.9 (18.7)
  30 minutes post-dose | 32.1 (21.5) | 33.4 (19.5)
  1 hour post-dose | 36.0 (24.3) | 34.0 (18.4)
  3 hours post-dose: number analyzed (Participants) | 9 | 5
  3 hours post-dose | 51.2 (23.4) | 48.4 (20.6)
  6 hours post-dose: number analyzed (Participants) | 9 | 4
  6 hours post-dose | 66.4 (25.1) | 69.3 (18.4)
  12 hours post-dose: number analyzed (Participants) | 9 | 4
  12 hours post-dose | 86.3 (25.0) | 78.0 (18.2)
  24 hours post-dose: number analyzed (Participants) | 9 | 5
  24 hours post-dose | 100.0 (36.5) | 93.8 (17.7)
  30 hours post-dose: number analyzed (Participants) | 9 | 5
  30 hours post-dose | 95.4 (32.6) | 90.6 (15.8)
  48 hours post-dose: number analyzed (Participants) | 9 | 5
  48 hours post-dose | 71.8 (29.1) | 79.2 (17.9)
  72 hours post-dose: number analyzed (Participants) | 9 | 5
  72 hours post-dose | 40.8 (37.8) | 44.6 (18.0)
  96 hours post-dose: number analyzed (Participants) | 9 | 4
  96 hours post-dose | 20.0 (23.5) | 16.0 (11.6)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study (approximately 32 months)
Arm/Group | Prior On-demand Participants | Switch Participants
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/13 | 2/10
Other Adverse Events (participants affected / at risk) | 10/13 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prior On-demand Participants (N=13) | Switch Participants (N=10)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prior On-demand Participants (N=13) | Switch Participants (N=10)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site irritation (General disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT02973087/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT02973087/SAP_001.pdf